CLINICAL TRIAL: NCT04681755
Title: Rehabilitation Required Due to Functional Neurological Impairment and Respiratory Disorders After Severe SARS-CoV-2 Infection in ICU Units
Brief Title: Rehabilitation Required Due to Clinical Disorders After Severe Covid-19 Infection
Acronym: REHABCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7725
Record Dates: First submitted 2020-12-21; First posted 2020-12-23 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Rehabilitation; SARS-CoV-2; COVID-19; Neurological function; Respiratory disorder; Intensive care unit
MeSH Terms: conditions — COVID-19; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the emergence of an epidemic cluster in Mulhouse, a city located 100 km south of Strasbourg, Alsace was one of the first French regions to be affected by the coronavirus (SARS-CoV-2 or COVID-19). As a result, all hospitals in the region, including both Strasbourg University Hospitals, had to deal with the epidemic wave earlier and more intensely than the rest of France. At the time of writing this article, 6 weeks after the start of the epidemic, we have counted 998 hospital deaths in our region, i.e., an intrahospital mortality rate linked to COVID-19 of 5.3 deaths per 10,000 inhabitants (https://dashboard.covid19.data.gouv.fr/).

Currently, our intensive care unit still has a large number of patients hospitalized for COVID-19. Some of these patients have severe damage to one or more organs, and in particular a neurological or respiratory deficit suggesting that they will need post-resuscitation rehabilitation. The primary aim is to assess the neurological disorder after severe SARS-CoV-2 infection and the second is the respiratory impairment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Patient hospitalized in surgical intensive care at the New Civil Hospital between February 24 and April 15, 2020.
* Patient with a SARS-CoV-2 infection documented by RT-PCR or with lesions suggestive on chest CT.
* Patient who has given his consent for the use of his data for the purposes of this research

Exclusion Criteria:

* Patient without documentation of SARS-CoV-2 infection (RT-PCR or chest scanner)
* Patient who expressed his opposition to participating in the study
* Subject under safeguard of justice
* Subject under guardianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with a SARS-CoV-2 infection documented by RT-PCR or with lesions suggestive on chest CT.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-05-19 (Estimated); Study Completion 2021-05-19 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of the neurological disorder after severe SARS-CoV-2 infection | The files analysed retrospectily from February 24, 2020 to April 15, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Strasbourg University Hospitals - Anesthesia and surgical resuscitation service, Strasbourg, France